CLINICAL TRIAL: NCT01618630
Title: Amino Acid Benefits in Pediatric Burn Patients Who Participate in Exercise.
Brief Title: Amino Acid Supplementation in Recovery From Severe Burns
Acronym: ExAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 12-048
Record Dates: First submitted 2012-05-30; First posted 2012-06-13 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Burn Injury
Keywords: burn injury; children; nutrition; lipid metabolism; insulin sensitivity; amino acids
MeSH Terms: conditions — Burns; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EAA Supplementation + Exercise Training (Experimental): Drink an amino acid supplementation during exercise training.
  Interventions: Dietary Supplement: EAA Supplementation + Exercise Training
- Placebo + Exercise Training (Placebo Comparator): Drink a placebo supplementation during exercise training.
  Interventions: Dietary Supplement: Placebo + Exercise Training

INTERVENTIONS:
Dietary Supplement: EAA Supplementation + Exercise Training — Amino acids in drinks between meals for exercise training period.
  Arms: EAA Supplementation + Exercise Training
Dietary Supplement: Placebo + Exercise Training — Placebo supplementation as drinks in between meals for exercise training period.
  Arms: Placebo + Exercise Training

SUMMARY:
Exercise during recovery is now Standard of Care at Shriners Hospital for Children Galveston, since positive effects of exercise training were found on lean body mass and recovery after burns. Essential amino acids (EAA) effective in healthy individuals.Thus, EAA supplementation in children recovering from burns, may potentially augment the effects of exercise by increase muscle mass, improve muscle fat oxidation, reduce tissue fat, and possibly improve insulin resistance.

DETAILED DESCRIPTION:
Severe burns result in persistent and extensive fat deposition in liver and muscle tissue. This may be related to the prolonged insulin resistance observed following burn. In this study the investigators will test the hypothesis that essential amino acids act in synergy with exercise to improve liver steatosis and muscle lipid metabolism, and thus also affect insulin sensitivity. Children with burns will participate in six weeks of exercise training with/without amino acid supplementation. Before and after the intervention, measurements will be done to determine muscle and liver fat content, muscle fat and protein metabolism, and insulin sensitivity.

We will prospectively enroll 40 children with ≥30% of their total body surface area (TBSA) burned. The age range will be 7-17 years. Children will be recruited from Shriners Hospitals for Children (SHC)-Galveston. Burned children will be randomized to undergo an exercise program in combination with daily intake of EAA (n=20) or a placebo drink (n=20). The exercise program and daily intake of AA will begin within the first week of discharge from the burn ICU (approximately 1-3 months post burn, when the patient's wounds are 95% healed). The definition of 95% healed is 7 days after the final autografting procedure. We anticipate enrolling 10 children per year for 4 years. Only children meeting the inclusion and exclusion criteria specified in the Human Subjects Section will be enrolled.

Nutritional Supplement: The nutritional supplement will be administered at a dose of 0.18 g/kg body weight of amino acids two times per day with the following composition: 3% histidine, 9% isoleucine, 36% leucine, 17% lysine, 4% methionine, 5% phenylalanine, 10% threonine, 7% valine, and 10% arginine. The dose and choice of amino acids is based on our preliminary data. Each dose is about 0.03 g/kg body weight higher than what has been shown effective in adults, as children have higher protein needs. We have shown that only EAA are needed to affect muscle protein synthesis and lean mass. Thus the amount given (g or kcal) can be restricted. As in our preliminary studies, we will include arginine in the EAA mixture, since arginine may have unique anabolic effects (55; 86). Placebo will consist of a mixture of inert components (sucralose and other pharmaceutical excipients). The supplement will be taken in two daily doses in the form of drinks (total daily dose of i.e., 0.30 g/kg body weight total per day), and intake recorded in a diary. The first dose will be taken between breakfast and lunch, and the second between lunch and dinner. For the children exercising before lunch, the first dose of EAA will be ingested immediately after exercise. Correspondingly, for children exercising after lunch, the second EAA dose of the day will be ingested immediately after exercise. If the child forgets to take one of the drinks during the day, he/she may take the second one between dinner and bedtime. During the weekends, parents/caregivers are instructed to take the dosage around the same time.

Data Analysis and Interpretation. To determine effects of amino acids on fat and muscle lipid stores, changes from pre- to post intervention in the two groups will be compared using ANCOVA. From the preliminary data, we expect that amino acids will decrease liver and plasma lipids.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 7-17 years old
3. Body weight >20 kg (based on blood requirements)
4. ≥30% Total Body Surface Area (TBSA)
5. Wounds 95% healed

Exclusion Criteria:

1. Respiratory insufficiency
2. Multiple fractures
3. History of Cancer in the last 5 years
4. Diabetes Mellitus
5. Bilirubin > 3 mg/dl
6. Associated head injuries requiring specific therapy
7. Associated injuries to chest or abdomen requiring surgery
8. Serum creatinine > 3 mg/dl after fluid resuscitation
9. Receipt of any experimental drug other than the ones supplied within two months of this study
10. Any metal in body including rods, cardiac defibrillator, pacemakers, etc
11. Orthopedic casting which would prevent placement of patient in MRI machine
12. Hepatitis
13. Abnormal EKG
14. Electrical burns
15. Patients unable to lie still without heavy sedation will be excluded from MRI portion.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2016-12-05 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Lean Muscle Mass | It is the change in time, from baseline until post exercise. Baseline is within the first week of discharge from the burn ICU, approximately 1-3 months post burn. Exercise training is 6-12 weeks.
  Is the total weight of your body minus all the weight due to your fat mass. It is measured in kilograms by dual X-ray absorptiometry scan.

SECONDARY OUTCOMES:
whole body lipolysis rate | It is the change in time, from baseline until post exercise. Baseline is within the first week of discharge from the burn ICU, approximately 1-3 months post burn. Exercise training is 6-12 weeks.
  A euglycemic-hyperinsulinemic clamp is performed over the last 2hr of the 4-hr isotope infusion. It is measured in μmol/kg body weight/min
Hepatic glucose release rate and whole body glucose uptake rate | It is the change in time, from baseline until post exercise. Baseline is within the first week of discharge from the burn ICU, approximately 1-3 months post burn. Exercise training is 6-12 weeks.
  A primed, constant (0.44 μmol/kg/min) infusion of [6,6-2H2]-glucose is used for glucose kinetics. A euglycemic-hyperinsulinemic clamp is performed over the last 2h of the 4-hr isotope infusion.It is measured in μmol/kg body weight/min.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar E Suman, PhD, Principal Investigator — UTMB, Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Galveston, Texas, United States